CLINICAL TRIAL: NCT00980759
Title: A Phase II Randomized Study of Prophylactic Irradiation of the Para-Aortic Lymph Nodes by 3-D Conformal Radiotherapy Technique With Concurrent Chemotherapy Based on the Hypoxic Status of Locally Advanced Uterine Cervical Cancer
Brief Title: Prophylactic Irradiation of the Para-Aortic Lymph Nodes in Locally Advanced Uterine Cervical Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Joo-Young Kim, Principal Investigator, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-209
Record Dates: First submitted 2009-09-18; First posted 2009-09-21 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Cervical Cancer
Keywords: Extended-field Irradiation (EFI); Cervical cancer; Hypoxia; Carbonic anhydrase 9 (CA9); locally advanced uterine cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Hypoxia

STUDY DESIGN:
Intervention Model Description: Randomization of Radiotherapy field
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EFI(Extended-Field Irradiation) (Experimental): Para-aortic and Pelvic Irradiation with chemotherapy(cisplatin)
  Interventions: Radiation: EFI
- Pelvic RT (Experimental): Pelvic Irradiation with chemotherapy(cisplatin)
  Interventions: Radiation: Pelvic RT

INTERVENTIONS:
Radiation: EFI — Para-aortic and Pelvic Irradiation with chemotherapy(cisplatin)
  Other Names: Extended-field Irradiation
  Arms: EFI(Extended-Field Irradiation)
Radiation: Pelvic RT — Only Pelvic Irradiation with chemotherapy(cisplatin)
  Other Names: Pelvic only treatment
  Arms: Pelvic RT

SUMMARY:
This study is an open-label, multi-institutional, randomized phase II study, which is designed to investigate the efficacy of Extended-field irradiation (EFI) on reducing recurrences at the para-aortic lymph node (PAN), and also on improving disease-free survival of locally advanced uterine cervical cancer. Radiotherapy is given as a conformal technique based on the individually taken CT scan and cisplatin is given concomitantly with radiotherapy in both EFI arm and pelvis only treatment arm. According to our past study result, patients with more hypoxic tumors are more likely to develop distant metastasis including the recurrences at PAN (1-3). This study started with examination of CA9 (hypoxia marker) expression in the primary cervical tumor before randomization because it was expected that there would be a differential benefit of EFI in patients with CA9-positive vs CA9-negative tumors. However, the study design was modified because there was too much delay in the patient with CA9-negative tumors. The patients are now registered and then immediately randomized to experimental (EFI) and control arm (pelvis only treated) with examination of CA9 expression at later time.

DETAILED DESCRIPTION:
Patients with primary, untreated, histologically confirmed carcinoma of the uterine cervix are included in this study. Absence of metastatic para-aortic lymphadenopathy is the prerequisite of the enrollment, and this is confirmed by imaging studies such as MRI covering the abdomen and pelvis, and PET/CT scan. The sample size is based on the previous studies (1-3). Considering that the disease-free survival of the experimental arm (patients who are treated with prophylactic para-aortic LN irradiation) and those who are not treated is 82% vs 72% (preliminary analysis), with the alpha error of 5% and statistical power of 90% (one-sided), a total of 140 patients in each treatment arm is needed. With 10% of follow-up loss taken into account, the total number of patients will be 312. Above figures were calculated on the basis of 80% statistical power and 5% type I error rate. PAN is treated prophylactically in the experimental arm with 45Gy/25F/5week fractionation schedule. Pelvis is treated according to the individual institute's practice guideline. Boost treatment for any enlarged pelvic lymph node or residual cervical/ parametrial disease with conformal radiation technique are allowed. Intracavitary radiation is given via low-dose-rate or high-dose-rate brachytherapy technique. Weekly cisplatin is given to all patients, however, when the patient's physical condition does not allow cisplatin administration, it can be omitted. This should be taken into account in the final analysis. The stage and the presence of pelvic lymphadenopathy are two stratification factors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (who have been adequately clinically staged) with primary, untreated, histologically confirmed invasive squamous cell carcinoma, adenocarcinoma, or adenosquamous carcinoma of the uterine cervix, FIGO stage IB1 with pelvic lymph node metastasis, IB2, IIA(≥4cm in tumor size, or pelvic LN metastasis), IIB, IIIA, IIIB with only unilateral pelvic wall extension, and IVA
2. Patients with negative, para-aortic lymphadenopathy determined by pelvic MRI and/or PET/CT scan.
3. Patients with adequate bone marrow function: ANC greater than or equal to 1,500/ul, platelets greater than or equal to 100,000/ul at the beginning.
4. Patients with adequate renal function: creatinine equal to or less than 2.0 mg/dL.
5. Patients who have signed an approved informed consent and authorization
6. Patients who have met the pre-entry requirements specified in section 6.0.
7. Patients with ECOG Performance Status of 0, 1, 2 and Karnofsky Performance Scale of 100, 90, 80, 70, 60, 50
8. Age: 18≤age≤80

Exclusion Criteria:

1. Stage IIIb with bilateral pelvic wall extension and stage IVB lesions are not eligible.
2. Patients with histology other than squamous, adeno, adenosquamous cell carcinoma
3. Patients who have received prior radiotherapy of pelvis or total hysterectomy Patients who have diagnosis of other malignant tumors other than non- malignant melanoma skin cancer or stage I. II papillary, follicular thyroid cancer.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2006-07-28; Primary Completion 2019-11-30 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of the Extended-Field Irradiation on the recurrence rate in para-aortic lymph nodes and the disease-free survival rate of the patients with locally advanced uterine cervical cancer | 5 years

SECONDARY OUTCOMES:
To evaluate overall survival, toxicities and quality of life (QOL) of the patients treated by EFI compared to the control group of patients | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joo-young J Kim, M.D., Ph.D., Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
undecided